CLINICAL TRIAL: NCT00672633
Title: A Double Blind Randomized Controlled Trial of Lovaza in Adolescents With Mild to Moderately Elevated Triglycerides.
Brief Title: Trial of Lovaza in Adolescents With Mild to Moderately Elevated Triglycerides
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Very slow recruitment.
Sponsor: Boston Children's Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Voula Osganian, Physician Scientist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08010028
Record Dates: First submitted 2008-04-30; First posted 2008-05-06 (Estimated); Results first posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Hypertriglyceridemia
Keywords: Omega 3 Fatty Acids; Triglycerides; Lovaza; Trial
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Omacor; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A , Experimental (Experimental): Lovaza, 4 grams/day orally for 6 months
  Interventions: Drug: Lovaza
- Corn Oil Pill (Placebo Comparator): Corn Oil Pill, 4 pills/day orally for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lovaza — Lovaza , 4 grams/day orally for 6 months
  Arms: A , Experimental
Drug: Placebo — Corn Oil Pill, 4 pills/day orally for 6 months
  Other Names: Corn Oil Pill
  Arms: Corn Oil Pill

SUMMARY:
The investigators will conduct a randomized clinical trial to evaluate the efficacy of Lovaza (formerly known as Omacor) in reducing triglyceride levels in youth ages 10-19 years old whose baseline triglycerides range from 150 mg/dl to 1000 mg/dl. Seventy subjects will be recruited at baseline and randomized to the treatment condition, Lovaza 4 grams/day for 6 months or the control condition, a corn oil placebo, 4 tablets a day for 6 months. Participants in both the treatment and control groups will receive the standard of care, which is dietary advice to follow a low, refined carbohydrate and low saturated fat diet that emphasizes increasing intake of fruits and vegetables and eating 2 servings per week of fishes rich in omega-3 fatty acids, consistent with the American Heart Association recommendations. The primary outcome will be change in fasting triglycerides from baseline to 3 months. The investigators hypothesize that patients who receive LOVAZA will have significantly greater reductions in plasma triglyceride levels when compared to patients on placebo at 3 months.

DETAILED DESCRIPTION:
The investigators propose to conduct a placebo controlled, double blind, parallel group randomized trial to evaluate the efficacy of Lovaza (formerly known as Omacor) in reducing triglyceride levels in youth ages 10-19 years old whose baseline triglycerides range from150 mg/dl to 1000 mg/dl. Seventy subjects will be recruited at baseline and randomized to the treatment condition, Lovaza 4 grams/day for 6 months or the control condition, a corn oil placebo, 4 tablets a day for 6 months. Participants in both the treatment and control groups will receive the standard of care, which is dietary advice to follow a low, refined carbohydrate and low saturated fat diet that emphasizes increasing intake of fruits and vegetables and eating 2 servings per week of fishes rich in omega-3 fatty acids, consistent with the American Heart Association recommendations (Kris-Etherton, 2003). Subjects will be randomized to the treatment or control condition after a 4 week run-in period of dietary education and advice. The primary outcome will be change in fasting triglycerides from baseline to 3 months.

2.0 SPECIFIC AIMS

2.1 Primary Aim/Outcome

* To determine the efficacy of LOVAZA in reducing plasma triglyceride levels among adolescents, ages 12-19 years with mild to moderate hypertriglyceridemia. We hypothesize that patients who receive LOVAZA will have significantly greater reductions in plasma triglyceride levels when compared to patients on placebo at 3 months.

2.2 Secondary Aims/Outcome

* To determine whether the efficacy of LOVAZA varies with duration of treatment, 3 months versus 6 months.
* To determine the effects of LOVAZA on plasma HDL and LDL cholesterol at 3 months and 6 months.
* To determine the effects of LOVAZA on systolic and diastolic blood pressure at 3 months and 6 months.

2.3 Exploratory Aims

* To describe the effects of LOVAZA on vascular reactivity/endothelial function as measured by pulse amplitude at 3 months and 6 months.
* To describe the effects of LOVAZA on levels of biomarkers of inflammation as measured by C-Reactive Protein at 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10-19 years old
* Fasting Triglyceride levels of 150-1000 mg/dl at the screening and baseline visit
* Ability to swallow pills
* Informed consent from a parent or legal guardian of minors or adult subject
* Written assent from the adolescent to participate in the study
* English or Spanish speaking

Exclusion Criteria:

* Food Allergy to Fish or any components of the pills which includes alpha tocopherol, partially hydrogenated vegetable oils including soybean oils and gelatin and glycerol or corn oil, and iron oxide or iron oxide containing food color additives.
* Pregnancy or positive urine pregnancy test for those females who have begun menstruating
* Breast feeding
* Alcohol Use: Patient is unable to abstain from alcohol use during the study. This will be assessed by asking the following questions: "During the past 30 days, on how many days did you have at least one drink of alcohol?"; "During the past 30 days, on how many days did you have 5 or more drinks of alcohol in a row, that is, within a couple of hours?"; "This study requires that you abstain from alcohol use during the course of the study. Do you think you can do this?"
* Known Bleeding Disorder or Coagulopathy or treatment with anticoagulant medications or low platelet counts, abnormal PT, or PTT.
* Significant cognitive or psychosocial disorder or medical illness that would limit participation in the trial.
* Type 1 or 2 Diabetes or fasting glucose that is >=126 mg/dl
* Liver disease or an ALT greater than 2 times upper limit of normal
* Treatment with medications that affect triglyceride levels, including oral hypoglycemic agents or insulin.
* Be currently taking the same oral contraceptive pills for less than the past three months or intend to change or discontinue prescription oral contraceptive pills used in the next seven months
* Be currently taking any over-the-counter supplements that affect triglycerides or lipid metabolism including over the counter fish oil supplements.
* Treatment for or diagnosis of a thyroid disorder or an elevated TSH level at baseline

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2008-04; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stavroula K Osganian, MD, ScD, Principal Investigator — Boston Children's Hospital; Sara DeFerranti, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recuited from medical clinics at Boston Children's Hospital and referrals from community pediatricians. Recruitment took place from July 2008 to October 2011.
Pre-assignment Details: Eligible patients participated in a 4 week dietary counseling run-in period before randomization. Patients were randomized if their triglycerides remained at or above 150 mg/dl after the 4 week run in period.
Groups:
- Lovaza: Treatment Arm: 4 grams/day orally for 6 months
- Placebo: Corn oil placebo: 4 pills/day orally for 6 months
Period: Overall Study
Arm/Group | Lovaza | Placebo
Started | 12 | 13
Completed | 12 | 12
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lovaza: Treatment Arm
- Placebo: Corn oil placebo
- Total: Total of all reporting groups
Arm/Group | Lovaza | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 12 | 23
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 13.3 (2.4) | 14.7 (2.7) | 14.0 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 5 | 9 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Triglycerides [Mean (Standard Deviation); unit: mg/dl] — Fasting Triglycerides
  mg/dl | 230 (44) | 225 (55) | 227 (49)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Triglycerides
Description: Fasting Triglycerides
Time Frame: 3 months
Population: Intention to Treat
Measure: Geometric Mean (Standard Error); unit: mg/dL
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | 171 (18) | 186 (20)
Statistical Analysis 1: Comparison: Lovaza vs Placebo; The study was designed with 80% power to detect a net improvement of Triglyceride elevles with a sample size of 60; Test type: Superiority or Other; p = 0.52, ANOVA; Repeated measures; Mean Difference (Net) = 20

2. Secondary Outcome: LDL Cholesterol
Description: Low Density Lipoprotein Cholesterol
Time Frame: 3 months
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | 116 (11) | 104 (11)
Statistical Analysis 1: Comparison: Lovaza vs Placebo; No power calculations done for this outcomes; Test type: Superiority or Other; p = 0.06, ANOVA; Repeated Measures; Mean Difference (Net) = 16

3. Secondary Outcome: HDL Cholesterol
Description: High Density Lipoprotein Cholesterol
Time Frame: 3 months
Population: Intention to Treat
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | 35.8 (1.7) | 33.6 (1.7)
Statistical Analysis 1: Comparison: Lovaza vs Placebo; No power calculations were conducted for this outcome; Test type: Superiority or Other; p = 0.27, ANOVA; Repeated Measures; Mean Difference (Net) = 2.3

ADVERSE EVENTS:
Arm/Group | Lovaza | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No